CLINICAL TRIAL: NCT06902909
Title: Laparoscopic Pectopexy and Laparoscopic Colporrhaphies in Pelvic Organ Prolapse Treatment
Status: Enrolling by invitation | Type: Observational
Sponsor: Tampere University Hospital (Other)
Collaborators: Seinajoki Central Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: R23076
Record Dates: First submitted 2025-03-17; First posted 2025-03-30 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: Vaginal Vault Prolapse; Uterine Prolapse; Cystocele, Midline; Rectocele; Female
Keywords: laparoscopic pectopexy; laparoscopic colporraphy
MeSH Terms: conditions — Pelvic Organ Prolapse; Uterine Prolapse; Cystocele; Rectocele

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Laparoscopic pectopexy with or without concomitant laparoscopic colporraphy: Patients undergoing laparoscopic pectopexy for pelvic organ prolapse, with or without concomitant laparoscopic anterior and posterior vaginal wall repair using sutures. The procedure involves the placement of a 3x15 cm Dynamesh PRP PVDF mesh to the vaginal apex or uterine cervical stump with monofilament and multifilament sutures and anchored to the pectineal ligaments bilaterally. Follow-up assessments will be conducted 12 months postoperatively to evaluate symptom relief, anatomical correction, and surgical safety.

SUMMARY:
This prospective cohort study investigates the surgical outcomes of laparoscopic pectopexy and laparoscopic colporraphy performed at the Wellbeing Services County of South Ostrobothnia. The primary outcome measure is to assess changes in sensation of bulge and pressure. Secondary outcome measures include evaluating other prolapse symptoms and pain, quality of life, anatomical correction of prolapse, surgical safety parameters, and postoperative complications. Approximately 40-50 laparoscopic pectopexies will be performed over two years by a single experienced surgeon. The study requires preoperative and postoperative assessments, including standardized patient questionnaires and anatomical measurements.

DETAILED DESCRIPTION:
The study aims to evaluate the effects of laparoscopic pectopexy and colporraphy on pelvic organ prolapse (POP) symptoms, anatomical prolapse repair, and surgical outcomes. The primary outcome measure is the presence of a bulging sensation 12 months after surgery. Secondary outcome measure includes additional prolapse-related symptoms, residual urine volume, pelvic pain, urinary incontinence, and safety parameters such as intraoperative blood loss and complications. Anatomical correction will be assessed using the Pelvic Organ Prolapse Quantification (POP-Q) system.

All surgical procedures will be performed by a single experienced surgeon with over five years of experience and more than 100 laparoscopic pectopexies performed. Patients will undergo laparoscopic pectopexy, with or without concomitant anterior and posterior vaginal wall repair using sutures. The pectopexy procedure utilizes a 3x15 cm Dynamesh PRP PVDF mesh, secured with absorbable monofilament thread to the vaginal cuff or with non-absorbable multifilament sutures to the uterine cervical stump.

ELIGIBILITY:
Inclusion Criteria:

* Symptomatic pelvic organ prolapse
* Uterine or vaginal vault prolapse reaching the hymenal ring (POP-Q classification: ≥0 cm)
* If uterus in situ, consent for supracervical hysterectomy
* Suitable for laparoscopic mesh surgery
* Age: 18-79 years
* Non-pregnant, no pregnancy desire.
* Sufficient Finnish language skills
* Concurrent anterior and/or posterior prolapse repair if POP-Q criteria met: tvl >8 cm and Aa, Ba, Ap, Bp ≥0

Exclusion Criteria:

* Unwillingness to undergo surgery or mesh implantation
* High anesthetic or surgical risk due to comorbidities
* Indication for laparoscopic sacrocolporectopexy due to rectal intussusception
* Desire to preserve the uterus
* Pregnancy or planning future pregnancy
* Inability to understand Finnish or study-related forms due to cognitive impairments
* Need for concomitant urinary incontinence surgery

Ages: 18 Years to 79 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Laparoscopic pectopexy and colporrhaphies are gynecological surgeries and are therefore exclusively offered to patients who are female by birth.
Study Population: Patients with symptomatic vaginal or uterine prolapse at least to the hymenal level and who have an indication for vaginal apex (DeLancey level I) prolapse repair using mesh are being recruited for the surgery.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2024-02-01 (Actual); Primary Completion 2027-02-28 (Estimated); Study Completion 2027-02-28 (Estimated)

PRIMARY OUTCOMES:
Patient-reported postoperative sensation of bulging at 12 months postoperatively | From the enrollment til follow-up visit at 12 months postoperatively
  During the history-taking process, symptoms such as a sensation of bulging or pressure are actively inquired about and documented accordingly. Results variables are presented as counts and percentages.

SECONDARY OUTCOMES:
Change in Pelvic Floor Organ function (PFDI-20 score) | From enrollment til the follow-up visit 12 months postoperatively
  Patients are asked preoperatively and postoperatively to complete the Pelvic Floor Distress Inventory (PFDI-20) that contains 4 different scores: POPDI-6, CRADI-8, UDI-6 and PFDI-20 Sum score. For statistical analysis about measurement score changes, paired t-test will be used. The differences are considered to be statistically significant at p-value of <0.05.
Change in sexual function and urinary incontinence (PISQ-12 score). | From the enrollment til follow-up visit at 12 months postoperatively
  Patients are asked preoperatively and postoperatively to complete the Pelvic Organ Prolapse/Urinary Incontinence Sexual Questionnaire (PISQ-12). For statistical analysis about measurement score change, paired t-test will be used. The differences are considered to be statistically significant at p-value of <0.05.
Change in quality of life. (15D questionnaire score) | From the enrollment til follow-up visit at 12 months postoperatively
  Patients are asked preoperatively and postoperatively to complete the Quality of Life 15D questionnaire. For statistical analysis about measurement score changes, paired t-test will be used. The differences are considered to be statistically significant at p-value of <0.05.
Change in pelvic pain (VAS score) | From the enrollment til follow-up visit at 12 months postoperatively
  Patients are asked to self-complete the Visual Analogue Scale (VAS) for pelvic pain both preoperatively and postoperatively. They are instructed to mark a cross or vertical line on a horizontal line labeled only with the endpoints: 0 (no pain) and 10 (worst possible pain), with no other numbers visible. A special ruler is used to determine the exact score based on the position of the mark, with results recorded to the nearest 0.5 points. For statistical analysis of changes in VAS scores, a paired t-test will be used. Differences will be considered statistically significant at a p-value of <0.05.
Post voiding residual in ml. | From enrollment til the follow-up visit 12 months postoperatively
  Postvoid residual (PVR) is measured by ultrasound during a transvaginal gynecological examination. Two dimensions are measured in centimeters in the sagittal plane, while the third dimension is consistently set at 10 cm. The PVR volume (in cubic centimeters) is calculated using the ellipsoid formula: a(cm)× b(cm) × c(10cm) × 0.52. One cubic centimeter is considered equivalent to one milliliter. For statistical analysis of changes in PVR measurements, a paired t-test will be used. Differences will be considered statistically significant at a p-value of <0.05.
Duration of surgery in minutes | From the beginning of surgery til the end of surgery
  During surgery, the following time measurements are recorded: total operative time (in minutes), defined as the duration from skin incision to completion of skin closure; and procedure-specific time (in minutes), which includes the time required for dissection of the pectopexy area, mesh application, and colporrhaphies. The results will be presented as the mean duration ± standard deviation (in minutes) and illustrated in a figure, with the X-axis representing individual cases and the Y-axis representing time in minutes for both types of measurements.
Estimated blood loss in ml | From the beginning of surgery til the end of surgery.
  Estimated blood loss during surgery will be recorded in milliliters (ml). The results will be presented as the mean ± standard deviation in ml.
Surgical Complications according to Clavien-Dindo classification. | From the beginning of surgery til 30 days postoperatively
  Surgical complications are recorded according to the Clavien-Dindo classification, from the beginning of surgery until 30 days postoperatively. Each adverse event is classified based on the Clavien-Dindo grading system. The results will be presented as counts and percentages of the study population in a table, where each complication is listed in a separate row and each grade of the Clavien-Dindo classification is represented in a separate column.
Hospitalisation duration in days | From the hospitalisation for surgery til discharge home.
  The duration of hospitalization is recorded in days, calculated from the hospitalisation for surgery until the day of discharge. The results will be presented as the mean ± standard deviation (in days).
Anatomical correction of prolapse according POP-Q classification | Right before the operaton til follow-up visit at 12 months postoperatively
  Anatomical correction is assessed during gynecological examination using the POP-Q system, both preoperatively and at the 12-month follow-up. The following points are measured: GH, PB, TVL, Aa, Ba, C, D, Ap, and Bp. For statistical analysis of changes in these measurements, a paired t-test will be used. Differences will be considered statistically significant at a p-value of <0.05.
Global impression of improvement. (PGI-I questionnaire) | At follow-up visit 12 months postoperatively
  Patient global impression of improvement (PGI-I) questionnaire is asked to fulfill by follow-up visit. It contains one question and seven answers. The results will be presented as counts and percentage for each possible answer.
Re-operation rate due to recurrence of vaginal apical prolapse, cystocele or rectocele. | From the end of surgery til follow-up visit at 12 months postoperatively
  The re-operation rate due to recurrence of vaginal apical prolapse, cystocele, rectocele will be recorded. Results will be presented as the number and percentage of patients requiring re-operation during the follow-up period.

CONTACTS AND LOCATIONS:
Overall Officials: Kirsi Kuismanen, MD, PhD, Study Chair — Tampere University; Kari Nieminen, MD, PhD, Study Chair — Tampere University
Locations (1):
- The Wellbeing Services County of South Ostrobothnia, Seinäjoki, Finland

IPD SHARING:
Plan to Share IPD: No
In this study, it is not possible to share IPD, because of several issues:
  1. Regulatory and Ethical Constraints: IPD will not be shared due to ethical considerations and data privacy regulations, including compliance with GDPR and other applicable laws protecting patient confidentiality.
  2. Lack of Consent for Data Sharing: participants did not provide explicit consent for data sharing beyond the primary study objectives.
  3. Institutional or Sponsor Policy: The study sponsor and institutional policies do not allow the sharing of individual participant data.
  4. Confidentiality and Privacy Risks: Due to the sensitive nature of the collected data and the risk of re-identification, IPD will not be made publicly available.
  5. No Plan for Secondary Use of Data: There are no current plans for sharing IPD as the study was not designed for secondary data use.